CLINICAL TRIAL: NCT04657874
Title: Association Between Bromelain and Escin in the Reduction of Postoperative Sequelae in Periodontal and Implant Surgery: Randomized Clinical Trial, Placebo-controlled, Double-blind
Brief Title: Bromelain and Escin in the Reduction of Postoperative Sequelae in Periodontal and Implant Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Collaborators: Dr. Leonardo Mancini (Unknown); Tommaso Pizzolante (Unknown)
Responsible Party: Principal Investigator, Enrico Marchetti, Prof. Enrico Marchetti, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RCT 002/2017
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain; Edema; Swelling Lips & Face
MeSH Terms: conditions — Pain, Postoperative; Edema; Facies | interventions — Bromelains; Escin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple blind randomization and computer-based random allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bromelain and Escin (Active Comparator)
  Interventions: Other: Bromelains and Escin Oral Tablet
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Bromelains and Escin Oral Tablet — Supportive care after oral surgery
  Other Names: Noflogo®
  Arms: Bromelain and Escin
Other: Placebo — Oral tablet without the active principle
  Arms: Placebo

SUMMARY:
A randomized clinical trial will be performed in parallel, placebo controlled, triple-blind to evaluate the effectiveness of the association Bromelina and Horse-chestnut (titrated in escin) (Noflogo®, Mavenpharma s.r.l., Rome, Italy) in the management of post trauma-surgery following surgery periodontal and implant surgery.

DETAILED DESCRIPTION:
At least 50 volunteers between the ages of 18 and 50, will be enlisted, with the need to perform one of the interventions described above and that fall within the criteria of inclusion.

The study will be carried out in accordance with the Helsinki Declaration on In Vivo Studies and will be initiated with the approval of the Internal Review Board of the University of L'Aquila.

The protocol follows the guidelines of the CONSORT Statement for parallel studies and will be recorded on the data base clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* No signs of gingival inflammation;
* FMBS and FMPS ≤ 20% after non-surgical causal therapy (Only for patients undergoing periodontal surgery)
* Smokers have to indicate how many cigarettes they smoke and how long have they been smoking

Exclusion Criteria:

* Gingival inflammation
* Positive anamensis for relevant systemic pathologies (renal, cardiovascular, hepatic, infectious, neoplastic and diabetological)
* Treatment with anti-inflammatory and/or antibiotics in the two weeks preceding the start of the trial
* History of allergy to one or more components of the medication to be tested
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Edema - Cheek Volume | Baseline
  The distance between the angle of the mouth and the lobe of the ear and the distance between the outer side of the eye and the angle of the jaw, following the bulge of the cheek. In addition, where possible, a facial scanner has been used.
Edema - Cheek Volume | Post-surgical - 30 min
  The distance between the angle of the mouth and the lobe of the ear and the distance between the outer side of the eye and the angle of the jaw, following the bulge of the cheek. In addition, where possible, a facial scanner has been used.
Edema - Cheek Volume | 2 days
  The distance between the angle of the mouth and the lobe of the ear and the distance between the outer side of the eye and the angle of the jaw, following the bulge of the cheek. In addition, where possible, a facial scanner has been used.
Edema - Cheek Volume | 7 days
  The distance between the angle of the mouth and the lobe of the ear and the distance between the outer side of the eye and the angle of the jaw, following the bulge of the cheek. In addition, where possible, a facial scanner has been used.
Trismus - Vertical Opening | Baseline
  A calibre has been used to measure vertical opening.
Trismus - Vertical Opening | Post-surgical - 30 min
  A calibre has been used to measure vertical opening.
Trismus - Vertical Opening | 2 days
  A calibre has been used to measure vertical opening.
Trismus - Vertical Opening | 7 days
  A calibre has been used to measure vertical opening.
Pain - (VAS) | Baseline
  The patient fills in the visual analog scale. This scale has values from 0 to 10 where 0 indicates "no pain" and 10 indicates "worst pain imaginable"
Pain - (VAS) | Post-surgical - 30 min
  The patient fills in the visual analog scale. This scale has values from 0 to 10 where 0 indicates "no pain" and 10 indicates "worst pain imaginable"
Pain - (VAS) | 2 days
  The patient fills in the visual analog scale. This scale has values from 0 to 10 where 0 indicates "no pain" and 10 indicates "worst pain imaginable"
Pain - (VAS) | 7 days
  The patient fills in the visual analog scale. This scale has values from 0 to 10 where 0 indicates "no pain" and 10 indicates "worst pain imaginable"

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, Division of Periodontology, L’Aquila, AQ, Italy

IPD SHARING:
Plan to Share IPD: Undecided